CLINICAL TRIAL: NCT04777695
Title: Sound Levels in the Pediatric Cardiac Critical Care Unit and Their Correlation With Sedation Administration, Delirium Scores and Patient Heart Rate
Status: Completed | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00013873
Record Dates: First submitted 2021-02-22; First posted 2021-03-02 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Noise Exposure; Sedative Withdrawal Delirium; Sedative Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CICU Inpatients: This is a prospective observational study of all children admitted to the pediatric CICU during a one month period of time for patients aged 0 to less than or equal to 22 years of age, as per the World Health Organization definition of a pediatric patient.
  Interventions: Other: Decibel Monitor

INTERVENTIONS:
Other: Decibel Monitor — Placement of a TeckPro data logging sound decibel meter at all patient bed-spaces to measure concurrent sound levels 24 hours per day, over a one (1) month period. Peak and mean sound levels per hour will be collected by the decibel monitor. Sound collected every 5 minutes will be logged by the decibel monitor and downloaded onto manufacturer software daily; data will then be imported into Microsoft Excel for further data analysis.

SUMMARY:
There is limited data regarding sound levels and burden in the pediatric cardiac critical care unit and how this compares with WHO standards. We seek to record this data and correlate sound level with bolus sedation administration, patient delirium scores, and patient heart rate trends.

Primary Outcomes

* 1 peak sound level in cardiac ICU in decibels
* 2 Mean sound level in cardiac ICU in decibels
* 3 Compare sound levels to WHO recommendations

Secondary Outcomes

* 1 To explore patient and unit factors that might influence these levels
* 2 To analyze sound levels in post-operative neonates, versus infants, versus children
* 3 To analyze patients on invasive versus non-invasine versus no ventilation

DETAILED DESCRIPTION:
This study aims to measure and average sound levels during hospitalization in the Children's National Pediatric Cardiac Intensive Care Unit (CICU) and investigate any correlation between heightened sound levels, the incidence of delirium, the administration of sedation medications given for agitation, and patient heart rate changes. Recognition of modifiable risk factors, such as sound levels, can lead to the development of preventive strategies to keep sound levels within recommended guidelines and to lessen the amount of sedation medications that are given for agitation. Successful completion of this research will contribute to the development of modifiable environmental factors for the prevention of oversedation and delirium in critically ill children, potentially improving outcomes in a vulnerable patient population. This will be the first study of this nature performed in a large CICU and the first to look at delirium scores and vital sign changes as related to sound levels.

Many studies have shown that increased sound levels in hospitals can worsen patient agitation and lead to sleep disturbance and impair rest and healing. The World Health Organization and the Environmental Protection Agency mandate that hospital sound levels not exceed 40-45 decibels dB(A) during the day and 35 dB(A) at night. Previous studies in four European ICUs with adult patients showed that ICUs demonstrated higher than recommended sound levels 50% of the time, with an average sound level of 51 dB(A) over 24 hours and a peak sound level of 85 dB(A). In the only published study on sound levels in a pediatric CICU and their relationship to sedation administration, Guerra et al showed in 2017 that mean levels were over 59dB in both open patient areas as well as single rooms with little variation between day and night levels and that a higher peak and average sound level correlated with more sedation boluses in the subsequent 2 and 5 hours respectively.

The association between neurotoxicity and the use of sedatives and analgesia in young infants with congenital heart disease has also been described. In addition, there are appreciable negative hemodynamic effects of oversedation on the pediatric patient recovering from cardiac surgery. For this reason, it is important to investigate the impact that sound levels might have on sedation administration. Along with this, as vital sign changes such as an elevated heart rate can lead to patients receiving additional sedation, it is equally important to study the relationship between patient heart rate and sound level in a cardiac intensive care unit.

Delirium is defined as an acute and fluctuating change in attention, thinking, perception, and consciousness secondary to an underlying medical condition. The consequences of delirium have been well studied in the adult critical care population, and include prolonged hospitalization time, difficulty with long-term thinking, increased days of mechanical ventilation, and increased risk of death after discharge from the hospital. In adult intensive care units, delirium screening is routinely performed because of the known consequences of the disease. With the advent of the Cornell Assessment of Pediatric Delirium (CAPD), there is now a rapid and reliable method of screening for delirium in pediatric intensive care units. Since 2018, bedside nurses in the Children's National CICU have been trained to calculate CAP-D scores. This delirium assessment performed once per shift, can be analyzed side-by-side with average sound levels over that same shift to assess for any correlation between these two parameters.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted to the pediatric CICU during a one month period of time for patients aged 0 to less than or equal to 22 years of age, as per the World Health Organization definition of a pediatric patient.

Exclusion Criteria:

* None

Max Age: 22 Years | Sex: All
Age Groups: Child, Adult
Study Population: Cardiac Critical Care patients include patients admitted for evaluation of congenital heart disease, status post repair of that disease, arrhythmia or for other management of pediatric patients with these conditions.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
To measure peak and mean sound levels in a cardiac ICU as well as sound dose and to compare this exposure to WHO recommendations | 1 month

SECONDARY OUTCOMES:
To correlate sound levels and sound dose with bolus sedation administered to these patients | 1 month
To correlate sound levels and sound dose with delirium scores in these patients | 1 month
To correlate sound levels and sound dose with patient heart rate | 1 month

OTHER OUTCOMES:
To explore patient and unit factors that might influence these levels a. To analyze sound levels in post-operative neonates, versus infants, versus children b. To analyze patients on invasive versus non-invasine versus no ventilation | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Yurasek, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garcia Guerra G, Joffe AR, Sheppard C, Pugh J, Moez EK, Dinu IA, Jou H, Hartling L, Vohra S; SedationWithdrawal and Analgesia Team (SWAT); Canadian Critical Care Trials Group (CCCTG). Prospective cohort study on noise levels in a pediatric cardiac intensive care unit. J Crit Care. 2018 Apr;44:318-322. doi: 10.1016/j.jcrc.2017.12.008. Epub 2017 Dec 14. PMID 29274594